CLINICAL TRIAL: NCT01546493
Title: Femoroacetabular Impingement: Correlating Hip Morphology to Changes in Cartilage and Subchondral Bone
Brief Title: Hip Impingement - Understanding Cartilage Damage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2009537
Record Dates: First submitted 2010-08-19; First posted 2012-03-07 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Controls (Experimental): Asymptomatic control subjects with no deformity. All patients will undergo all 3 interventions: MRI, qCT, and motion analysis.
  Interventions: Radiation: MRI; Radiation: qCT; Other: Motion Analysis
- Symptomatics (Experimental): Subjects with bilateral cam deformity and unilateral symptoms. All patients will undergo all 3 interventions: MRI, qCT, and motion analysis. Select patients will be asked to participate in a PET-MRI scan being conducted at The Royal Ottawa.
  Interventions: Radiation: MRI; Radiation: qCT; Other: Motion Analysis; Radiation: PET-MRI
- Asymptomatic (Experimental): Asymptomatic subjects with cam deformity. All patients will undergo all 3 interventions: MRI, qCT, and motion analysis. Select patients will be asked to participate in a PET-MRI scan being conducted at The Royal Ottawa.
  Interventions: Radiation: MRI; Radiation: qCT; Other: Motion Analysis; Radiation: PET-MRI

INTERVENTIONS:
Radiation: MRI — MRI scan. 3.0 Tesla MRI scans of both hips using Tip(T1-rho) and ultra-short echo time (UTE) sequences.
Radiation: qCT — Quantitative computed tomography(QCT) scans using a CT phantom
Other: Motion Analysis — 3D motion analysis to assess hip function.
Radiation: PET-MRI — Positron emission tomography combined with magnetic resonance imaging (PET-MRI) is a technology that will help us examine bone and cartilage at the molecular level.
  Other Names: Positron emission tomography-magnetic resonance imaging
  Arms: Asymptomatic; Symptomatics

SUMMARY:
Femoro-acetabular impingement (FAI) is a known cause of hip pain and possibly a major cause of adult hip osteoarthritis. The relationship between cam-type FAI deformity characteristics and joint degradation to better identify 'at-risk' patients requiring corrective surgery will be scrutinized to gain a better understanding of the condition's natural history. The influence of certain morphologies (e.g. size and location of the deformity) will be analyzed to determine if this leads to aberrant loading of regions of the cartilage and subchondral bone, resulting in cartilage damage and joint degradation. Additionally, this research will determine if changes in the subchondral bone precede cartilage degeneration.

The methodology for establishing the morphology/cartilage degeneration relationship includes Magnetic Resonance Image (MRI) analysis, three-dimensional motion analysis and computer simulation/finite element analysis.

The outcomes of this research may lead to a reduction in total hip replacement cases by as much as 70%, saving many Canadians from a painful and debilitating condition and reducing costs to the Canadian health care system by as much as $290 million annually.

DETAILED DESCRIPTION:
The research objectives are:

1. To determine the factors of cam deformities, including morphological, functional and bone quality, that are associated with cartilage degeneration through shape analysis, kinematic analysis, MRI imaging and bone densitometry.
2. To determine whether subchondral bone changes occur before detectable cartilage degeneration by examining magnetic resonance images of asymptomatic subjects who have an identifiable deformity.
3. To use 3D motion and finite element analysis to examine differences in mechanical stimuli in the subchondral bone and cartilage that are associated with FAI, thus expanding our understanding of the pathomechanisms of associated degeneration.

Three subject cohorts will be recruited: subjects with bilateral cam deformity and unilateral symptoms (Group I, 'active cartilage damage stage'), asymptomatic subjects with cam deformity (Group II, 'early stage') and asymptomatic control subjects with no deformity (Group III).

ELIGIBILITY:
Inclusion Criteria:

* Group I: Subjects with bilateral cam deformity and unilateral symptoms; Hip pain longer than 6 months referred to the groin/lateral aspect of hip; Positive impingement sign (determined by the surgeon); Plain radiographs: absence of arthritis (Tonnis Grade 0 or 1), absence of dysplasia (center edge >25 degrees) on AP radiograph, α-angle greater than 55 degrees on the Dunn view.
* Group II: Asymptomatic subjects with cam deformity; These patients will be recruited from our prevalence study (2006.813) with 200 asymptomatic individuals using MRI with radial sequences.
* Group III: Asymptomatic control subjects with no deformity; These patients will be recruited from our prevalence study (2006.813) which established their hip joint as having a normal femoral head neck contour. These subjects will be age-matched to Group I.

Exclusion Criteria:

* Participants who do not meet the criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-08-04 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | 24 months
  Patients will undergo MRI modalities which are sensitive to biochemical markers (T1-rho) and bone porosity (ultra-short echo time [UTE]) to evaluate joint cartilage. The T1-rho imaging is used to detect early molecular and biochemical alterations to cartilage while the UTE imaging is used to assess bone porosity. MRI scans will be completely pre-operatively and at a minimum of 24 months post-operatively.

SECONDARY OUTCOMES:
Quantitative Computed Tomography (qCT) | 24 months
  Patients will undergo a CT scan of the hip (qCT) that is sensitive to the mineral content within bone tissue, and can assess bone mineral density, a strong predictor of bone strength and stiffness, which can influence the health of the cartilage. This scan will take approximately 15 minutes.
Quantitative Motion Analysis to assess hip joint function | 24 months
  Hip joint kinematics and contact forces will be analyzed in the same subjects undergoing imaging analysis to better understand the role of joint function in the degeneration process. Patients will have 16 pairs of surface electromyography (EMG) electrodes placed on certain area of the skin. The kinematic and kinetic data will be recorded for all 3 groups. Data will be recorded during normal level walking and during completion of simulated daily tasks (uphill, downhill walking, stairs, squatting, sitting, rising from a chair).
Positron emission tomography-magnetic resonance imaging (PET-MRI) | 24 months or greater after original enrolment
  Positron emission tomography combined with magnetic resonance imaging (PET-MRI) is a technology that will examine bone and cartilage at the molecular level.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Beaule, MD, FRCSC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada